CLINICAL TRIAL: NCT06099405
Title: The Impact of Yoga Training Protocols on Cognition, Aerobic, and Neuromuscular Performances, and Retinal Microvasculature and Microcirculation in Older Persons.
Brief Title: Yoga Training and Retinal Vasculature
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: McKnight Brain Research Foundation (Unknown)
Responsible Party: Principal Investigator, Joseph Signorile, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20230735
Record Dates: First submitted 2023-10-19; First posted 2023-10-25 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Cognitive Change

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-speed, Cognitive Challenge Yoga (Experimental): Participants in this group will receive high-speed yoga training for 24 consecutive weeks for a total of 72 training sessions.
  Interventions: Behavioral: High-speed, Cognitive Challenge Yoga
- Traditional Yoga (Active Comparator): Participants will perform standard Hatha yoga with slow controlled speed movements for 24 consecutive weeks for a total of 72 training sessions.
  Interventions: Behavioral: Traditional yoga

INTERVENTIONS:
Behavioral: High-speed, Cognitive Challenge Yoga — Participants in this group will receive high-speed yoga with cuing 3 times per week for 24 consecutive weeks for a total of 72 training sessions of 1 hour duration. Subjects will move as quickly as possible from one pose to another.
  Arms: High-speed, Cognitive Challenge Yoga
Behavioral: Traditional yoga — Participants will perform controlled speed Hatha yoga 3 times per week for 24 weeks for a total of 72 sessions of 1 hour duration.
  Arms: Traditional Yoga

SUMMARY:
This study will compare the impact of a novel high-speed, cued yoga program to a standard yoga program on retinal microvasculature, cognition and neuromuscular function.

ELIGIBILITY:
Inclusion Criteria:

1. 60-90 years of age;
2. Montreal Cognitive Assessment (MoCA) > 23
3. no memory loss complaints

Exclusion Criteria:

1. uncontrolled cardiovascular or neuromuscular diseases that prevent participation in a training program;
2. cerebrovascular disease;
3. documented HIV infection or other immunodeficiency syndrome;
4. any systemic inflammatory or autoimmune conditions such as rheumatoid arthritis, systemic lupus erythematosus, or other serious concomitant medical illness;
5. a history of ocular surgeries (except for cataract surgery more than 6 months ago) or other ocular diseases;
6. bilateral moderate or severe cataracts;
7. refractive errors of myopia, hyperopia and/or astigmatism more than 6.0 Diopters

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
Changes in Retinal measured in microliters per second (ul/s) | Baseline, 24 weeks
  Measurements of retinal blood flow (ul/s)
Changes in Retinal vascular biomarkers | Baseline, 24 weeks
  vessel density in unitless fractal dimension.
Changes in the Hopkins Verbal Learning Test | Baseline, 24 weeks
  The Hopkins Verbal Learning Test assesses immediate recall, delayed recall, and delayed recognition. It is administered by reading 12 words aloud, then asking the client to verbally repeat the list of words (immediately; then after a delay) and identify the words from a 24-word list that is presented verbally. The word list includes words from the previous list, words related to the previous list, and words unrelated to the list. Units of measurement are points. The test has three recall trials of 12 words each scored from 0 (none remembered to 12 (all remembered). Therefore, there are 36 points available for the 3 trials. After 20-25 minutes the subject's delayed recall is tested as the subject is asked to recall the same list of words, scored 0-12. Then a retention trial using a list of 24 words (12 words from the previous list, 6 related words, and 6 unrelated words) is read. The subjects must identify if each word was on the previous list or not.
Changes in Executive Function | Baseline, 24 weeks
  Changes in executive function age-corrected fluid cognition composite score measured by the Dimensional Change Card Sort test, the Flanker test, Picture Sequence Memory test, List Sorting test, and pattern comparison test of the NIH Toolbox Cognition Module. The units of measurement are points with higher scores indicating higher levels of functioning. Scores 70 or below indicates significant fluid cognitive impairment, scores around 85 indicate below average fluid cognitive ability, scores at or near 100 are considered average, scores around 115 are considered above-average fluid cognitive ability, and 130 and above indicate superior fluid cognitive ability (top 2% based on the national Toolbox normative data).
Changes in the Six-Minute Walk Test | Baseline, 24 weeks
  The object of the test is to walk as far as possible for six minutes. The subject will walk at a normal pace around a marked course for six minutes. The subject may stop to rest and begin again at will. The distance covered indicates aerobic fitness. The further a person walks, the better their cardiovascular condition. The units are meters.
Changes in the Timed Up and Go | Baseline, 24 weeks
  Upon verbal cue, the subject stands up, walks around a cone placed three meters from the front edge of the chair, and then returns to a seated position as quickly as possible. Time is measured in seconds. The faster the person completes the test the better the dynamic balance.
Changes in One repetition Maximum Strength | Baseline, 24 weeks
  A one-repetition maximum test measures the maximum load that an individual can lift only a single time throughout the full range of motion of the chest press and leg press exercises using proper form. All subjects' one repetition maximum values will be determined within four to five trials. The units of measure are kilograms. Testing is performed on computerized, pneumatic machines.
Changes in Neuromuscular Power Testing | Baseline, 24 weeks
  Peak muscle power is then measured at eight relative intensities (40, 50, 60, 70, and 80% of one repetition maximum) on the computerized, pneumatic machines. For each repetition, the concentric phase is performed as fast as possible, and the eccentric phase lasts between 2 and 3 seconds. Power testing is done for the leg press and chest press and the unit of measurement is Watts.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph F. Signorile, PhD, Principal Investigator — University of Miami
Locations (1):
- Laboratory of Neruomuscular Research and Active Aging, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: No